CLINICAL TRIAL: NCT06882876
Title: Phase Ib Exploratory Study on the Combination of JS014 and Toripalimab in Combination With Transarterial Chemoembolization for Unresectable Hepatocellular Carcinoma.
Brief Title: JS014 Combined With Toripalimab and TACE in Unresectable HCC: a Phase Ib Study
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS014-F01
Record Dates: First submitted 2024-11-21; First posted 2025-03-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: JS014; Toripalimab; BCLC Stage B Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JS014 combined With Toripalimab and TACE (Experimental)
  Interventions: Drug: JS014 Combined With Toripalimab and TACE

INTERVENTIONS:
Drug: JS014 Combined With Toripalimab and TACE — JS014 (60μg/kg,QW)+Toripalimab (240mg , Q3W)+ dTACE (60mg/m2)

SUMMARY:
This is an open-label, single-center, single-arm phase Ib clinical trial. The aim of this study is to assess the safety and efficacy of JS014 in combination with Toripalimab and transarterial chemoembolization (TACE) for unresectable hepatocellular carcinoma (HCC). The primary endpoint is the safety and tolerability, while the secondary endpoints include objective response rate (ORR), disease control rate (DCR), time to progression (TPP), progression-free survival (PFS), and overall survival (OS).

DETAILED DESCRIPTION:
There is already existing evidence indicating that the efficacy of PD-1/PD-L1 therapy is closely associated with the immune response status within the tumor microenvironment. Researchers are now embarking on exploring immune-activating treatment approaches that can synergize with immunotherapy in the battle against cancer. This includes local treatments such as radiation therapy and local ablation therapy, which can induce local inflammation and release antigens to activate anti-tumor immune responses and enhance the efficacy of PD-1 antibodies. Multiple preclinical studies have confirmed that transarterial chemoembolization (TACE) and radiofrequency ablation (RFA) can induce immunogenic necrosis and activate anti-tumor immune responses. This study is designed to investigate the safety and efficacy of TACE combined with JS014 and Toripalimab in the treatment of advanced liver cancer. It is an open-label, single-center, single-arm phase Ib clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form, voluntarily participate in this study, good compliance and follow-up cooperation.
* Histologically or pathologically confirmed unresectable hepatocellular carcinoma;
* Male or female patients aged 18-75 years;
* Eastern Cooperative Oncology Group (ECOG) PS score of 0-1;
* Child-Pugh score of ≤7;
* BCLC/B stage; not previously treated with anti-cancer therapy; at least one measurable lesion (according to RECIST 1.1 criteria).
* Sufficient organ function in vital organs (excluding serious functional impairment in the heart, lung, liver, kidney, bone marrow, nervous system, and endocrine systems).

Exclusion Criteria:

* Diagnosed with fibrolamellar carci-noma of liver, intrahepatic cholangiocarcinoma, and mixed carcinoma;
* Within 28 days prior to the start of the study, the participant received treatment with another investigational drug or participated in another clinical study for a different therapeutic indication.;
* Based on the investigator's judgment, the patient is expected to live for less than 12 weeks;
* Uncontrolled pleural effusion, pericardial effusion, or ascites of moderate volume or more;
* Current or past history of central nervous system metastasis;
* Have a history of psychotropic drug abuse or drug use;
* Hereditary or acquired tendency towards bleeding and thrombosis, a thromboembolic event occurred within the past 6 months;
* Have a history of severe allergy to any monoclonal antibody, Toripalimab , JS014 and other ingredients of this study;
* Pregnant or breastfeeding women;
* Subjects with other factors that, in the judgment of the investigator, may cause the study to be prematurely terminated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse events | Two years
  Safety and tolerability

SECONDARY OUTCOMES:
ORR (RECIST 1.1) | Two years
  Objective response rate
DCR | Two years
  disease control rate
PFS | Two years
  Progression free survival
TTP | Two years
  time to progress
OS | Two years
  Overall survival
ORR(mRECIST) | Two years
  Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Liangrong Shi, M.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided